CLINICAL TRIAL: NCT01876537
Title: Phase 1 STRENGTHENING OF THE SACROCOCCYGEAL FASCIA IN THE SURGICAL TREATMENT OF PILONIDAL SINUS DISEASE
Brief Title: Hardware Wound Healing In Surgical Treatment Of Sacrococcygeal Pilonidal Sinus Disease
Acronym: HWHPSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Voronezh N.N. Burdenko State Medical Academy (Other)
Responsible Party: Principal Investigator, Brezhnev Stanislav Gennadievich, Ph.D., Voronezh N.N. Burdenko State Medical Academy
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: ZHKB-2015
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Sacrococcygeal Pilonidal Sinus Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual surgery (Active Comparator)
  Interventions: Device: Usual Surgery
- Hardware wound healing (Active Comparator)
  Interventions: Device: Hardware wound healing

INTERVENTIONS:
Device: Hardware wound healing
  Arms: Hardware wound healing
Device: Usual Surgery
  Arms: Usual surgery

SUMMARY:
THEME RELEVANCE. Sacrococcygeal pilonidal sinus disease (SPD) is a congenital disease that's well spread and constitutes 1-2% of all surgical pathologies. In all Coloproctological pathologies, the disease composes 14-20% (G.I. Vorobjov, 2006; V.D. Fedorov, 2005; Gupta P.J. et al., 2005). Clinical manifestations of pilonidal sinus disease mainly due to the appearance of inflammation in it.

The main approach in the complex treatment of this group of patients is to execute radical surgery. The guiding principles in it are adequate sanation and drainage of purulent focus.

Despite the fact that this disease is the subject of numerous medical journals, monographs, research works, masters and doctoral theses, frequency of unsatisfactory outcomes remains high (recurrence - from 10% to 19%, wound inflammation - 20-30%). In this case terms of stationary and out-patient treatment increase till 30-70 days (G.I. Vorobjov, 2006; B.M. Dacenko et al., 2004; Cubukcu А., 2001, Perruchoud С, 2002).

The frequency of unsatisfactory results after excision of SPD directly depends on the kind of surgery. After palliative surgery (incision and drainage of abscess) in 11.7 - 25.2% of patients occurs recurrence of the disease (McCallum I., King P.M., Bruce J., 2007;), for the open wound healing recurrence occur in 3-8% of the operated. For primary wound healing in 7,5-9,7% required re-surgery (V.K. An, 2003; A.A. Kartashev, 2011).

Sacrococcygeal pilonidal sinus disease overwhelmingly affects people, mostly young working age, and treatment failure leads to long-term temporary disability of patients.

In the last few years continue to discuss methods of one-time or multi-stage radical surgical treatment of pilonidal sinus, but to date there is no single approach to the choice of surgical treatment for this disease (V.L. Denisenko, 2008).

Success of surgical treatment of SPD depends on the development and introduction of new devices and techniques exist to produce convergence and immobilization of the wound edges, thereby obtaining its primary healing and a significant reduction of wound surface.

The high frequency of the disease and postoperative complications, as well as long-term temporary disability of patients demonstrates the relevance of the development of modern methods of radical surgery of sacrococcygeal pilonidal sinus disease (V.I. Pomazkin, 2008).

AIM OF RESEARCH. The aim of our research is to improve the results of complex radical surgical treatment of patients of sacrococcygeal pilonidal sinus disease through the development and introduction of new devices and techniques for convergence and immobilization wound edges.

TASKS OF RESEARCH.

1. To conduct a comparative analysis the most common surgical treatment of SPD in the frequency of complications in the intra- and postoperative periods.
2. To develop a device for convergence and immobilization wound edges in patients with SPD.
3. To analyze the effectiveness of the developed techniques and devices in comparison with traditional surgical treatment.
4. To make practical recommendations on the options and methods of using the developed methods and devices.

NOVELTY OF RESEARCH. For the first time, based on the design and creation of an approximation-immobilization device (RU Patent № 112020, Bull. № 1, 01.10.2012) will be improved the surgical treatment of patients with this pathology, clinical and anatomical study of the proposed device for different configurations of gluteal-sacrococcygeal region, as well as the analysis and justification of the basic parameters of wound (length, depth and width of the wound, the number of stitches, the complication rate , the area of the wound).

Developed a method of closure of the wound defect after radical excision of pilonidal sinus by Krivonosov-Brezhnev (RU Patent № 2,464,943, Bull. № 30 from 10.27.12.), that significantly reduces the risk of postoperative complications in patients with acute inflammation of the SPD.

For the first time an analysis of postoperative period in patients operated with the proposed methods compared with traditional methods of surgery was performed.

POSSIBLE APPLICATION AREAS. Results of the research designed for use in the treatment process of coloproctological departments at all levels, as well as the learning process of medical schools.

EXPECTED EFFECTIVENESS.

1. Scientific and technical effect: developed new techniques and devices for convergence and immobilization wound edges used for the treatment patients with SPD.
2. Medical and social effects: the introduction into clinical practice of the developed techniques and devices will improve the results of surgical treatment of patients with SPD by rigid fixation of wound edges, by reducing the time of postoperative wound healing, by decreasing the risk of complications in the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Sacrococcygeal pilonidal sinus disease
* Must be able to transfer surgery
* Should not be allergic to antibiotics

Exclusion Criteria:

* Low blood coagulation
* Вiseases, reducing immunity
* Insanity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
primary wound closure | up to 10-15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Voronezh Regional Hospital #1, Voronezh, Voronezh Regional, Russia